CLINICAL TRIAL: NCT06093503
Title: Phase 3, Open-Label, Randomized, Controlled, Global Study of Telisotuzumab Vedotin (ABBV-399) Combined With Osimertinib vs Platinum-Based Chemotherapy in Subjects With c-Met Overexpressing (OE) EGFR Mutant, Locally Advanced/Metastatic Non-Squamous NSCLC After a First Progression on Prior Third Generation EGFR TKi Treatment
Brief Title: Study of Intravenous Telisotuzumab Vedotin in Combination Osimertinib or Standard of Care Chemotherapy to Assess Change in Disease Activity in Adult Participants With Non-Small Cell Lung Cancer That Has a Mutation in the Epidermal Growth Factor Receptor Gene and That Overexpresses the c-Met Protein
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M22-142; 2022-502283-20-00 (Other: EU CT)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Telisotuzumab Vedotin; ABBV-399; Osimertinib; Cisplatin; Carboplatin; Pemetrexed; c-Met; NSCLC; Teliso-V; TeliMET NSCLC-03
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — telisotuzumab vedotin; osimertinib; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telisotuzumab Vedotin and Osimertinib (Experimental): Participants will receive telisotuzumab vedotin every 2 weeks in combination with osimertinib, until disease progression or unacceptable toxicity.
  Interventions: Drug: Telisotuzumab Vedotin; Drug: Osimertinib
- Standard of Care (Experimental): Participants will receive standard of care chemotherapy (carboplatin/pemetrexed or cisplatin/pemetrexed as prescribed by the physician), until disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Telisotuzumab Vedotin — Intravenous (IV) Infusion
  Other Names: ABBV-399
  Arms: Telisotuzumab Vedotin and Osimertinib
Drug: Osimertinib — Oral: Tablet
  Arms: Telisotuzumab Vedotin and Osimertinib
Drug: Cisplatin — IV Infusion
  Arms: Standard of Care
Drug: Carboplatin — IV Infusion
  Arms: Standard of Care
Drug: Pemetrexed — IV Infusion
  Arms: Standard of Care

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. Non-small cell lung cancer (NSCLC) is a solid tumor, a disease in which cancer cells form in the tissues of the lung. The purpose of this study is to assess how telisotuzumab vedotin in combination with osimertinib affects the disease state compared to standard of care in adult participants with locally advanced/metastatic non-squamous NSCLC that has a mutation in the epidermal growth factor receptor (EGFR) gene and that overexpresses the c-Met protein. Change in disease activity will be assessed.

Telisotuzumab vedotin is an investigational drug being developed for the treatment of NSCLC that overexpresses the c-Met protein. Participants are randomly placed in one of the two groups to receive telisotuzumab vedotin and osimertinib or standard of care chemotherapy. Approximately 250 adult participants with locally advanced/metastatic non-squamous NSCLC that has a mutation in the EGFR gene and that overexpresses the c-Met protein will be enrolled in the study in approximately 180 sites worldwide.

Participants will receive intravenous telisotuzumab vedotin every 2 weeks in combination with oral osimertinib tablets daily or standard of care chemotherapy (carboplatin/pemetrexed or cisplatin/pemetrexed as prescribed by the physician). Overall duration of the study is estimated to be approximately 47 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must have metastatic/locally advanced non-squamous NSCLC with documented epidermal growth factor receptor (EGFR) mutation del19 or L858R, with or without T790M mutation, and no identified EGFR mutations known to confer resistance to osimertinib (for instance C797S).
* Must have c-Met overexpressing non-small cell lung cancer (NSCLC) as assessed by an AbbVie designated immunohistochemistry (IHC) laboratory.
* Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Must have measurable disease per response evaluation criteria in solid tumors (RECIST) version 1.1.
* Must have received one prior regimen in the metastatic setting, consisting of a third generation epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKi) (for instance, osimertinib). Participant must have had one disease progression while on this third generation EGFR TKi. Prior-rechallenge with a third generation EGFR TKi is not allowed. Treatment with a first or second generation EGFR TKi immediately prior to the third generation EGFR TKi will not count as one prior regimen. Those who have received a third generation EGFR TKi as adjuvant therapy, and have progressed within 6 months of the last dose of treatment will be eligible (i.e., considered as having received a third generation EGFR TKi in the metastatic setting).
* Must be considered appropriate for platinum therapy based on the assessment of the treating physician.
* Participants with metastases to the central nervous system (CNS) are eligible only after definitive therapy (such as surgery or radiotherapy) is provided and:

  * There is no evidence of progression of CNS metastases at least 4 weeks after definitive therapy.
  * Participant is asymptomatic and off or on a stable or reducing dose of systemic steroids and/or anticonvulsants for at least 4 weeks prior to first dose of telisotuzumab vedotin.
  * There is no leptomeningeal seeding of the disease.
* History of prior radiation pneumonitis in the radiation field (fibrosis) is permitted.

Exclusion Criteria:

* Have adenosquamous histology, nor sarcomatoid features.
* Alterations in ALK, ROS1, or BRAF that predict sensitivity to targeted therapies.
* Have small-cell histology.
* Have received prior chemotherapy in the metastatic setting. For the enrollment criterion, if a subject has received one to two cycles of platinum-based chemotherapy prior to starting a third generation EGFR TKi, without progression and while awaiting EGFR status results, it will not be counted as "prior platinum therapy." Those who have received platinum-based chemotherapy as adjuvant therapy, and have progressed within 6 months of the last dose will be counted as having received a prior platinum therapy in the metastatic setting.
* Have a history of other malignancies except those listed in the protocol.
* Have a history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Have unresolved adverse events (AEs) >= Grade 2 from prior anticancer therapy, except for alopecia or anemia.
* Have had major surgery within 21 days prior to the first dose of telisotuzumab vedotin.
* Have clinically significant condition(s) including but not limited to those listed in the protocol.
* Clinically significant liver disease, including hepatitis, current alcohol abuse, or cirrhosis.
* Grade >= 2 edema or lymphedema.
* Grade >= 2 ascites or pleural effusion.
* Grade >= 2 neuropathy.
* Active uncontrolled bacterial or viral infection.
* Active corneal disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2028-04-11 (Estimated); Study Completion 2028-04-11 (Estimated)

PRIMARY OUTCOMES:
PFS in the Population of Participants with no Central Nervous System (CNS) Metastases at Baseline | Up to Approximately 41 Months
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 per ICR or death from any cause, whichever occurs earlier. Participants with no PFS event will be censored at the last evaluable radiographic assessment per ICR. Participants with no event and no evaluable post-baseline assessment will be censored at randomization.

SECONDARY OUTCOMES:
PFS in the Overall Population | Up to Approximately 41 Months
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 per ICR or death from any cause, whichever occurs earlier.
Overall Response (OR) in the Population of Participants with no CNS Metastases at Baseline | Up to Approximately 41 Months
  OR (per ICR) is defined as participants achieving a best overall response of confirmed complete response (CR) or confirmed partial response (PR) per ICR based on RECIST v1.1.
OR in the Overall Population | Up to Approximately 41 Months
  OR (per ICR) is defined as participants achieving a best overall response of confirmed CR or confirmed PR per ICR based on RECIST v1.1.
Duration of Response (DoR) in the Population of Participants with no CNS Metastases at Baseline | Up to Approximately 41 Months
  DoR is defined for confirmed responders as the time from the initial response (CR or PR) per ICR to the first occurrence of radiographic progression per RECIST v1.1 or death from any cause, whichever occurs first.
DoR in the Overall Population | Up to Approximately 41 Months
  DoR is defined for confirmed responders as the time from the initial response (CR or PR) per ICR to the first occurrence of radiographic progression per RECIST v1.1 or death from any cause, whichever occurs first.
Overall Survival (OS) in the Population of Participants with no CNS Metastases at Baseline | Up to Approximately 41 Months
  OS is defined as the time from randomization to the event of death from any cause.
OS in the Overall Population | Up to Approximately 41 Months
  OS is defined as the time from randomization to the event of death from any cause.
Change in Physical Functioning using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module 13 (EORTC QLQ-LC13) in the Population of Participants with no CNS Metastases at Baseline | Up to 41 Months
  The EORTC QLQ-LC13 is the lung cancer specific module of the core EORTC QLQ-C30.2 The QLQ-LC13 includes 13 questions that include both multi-item and single-item scales of lung cancer-associated symptoms (e.g., pain, coughing, hemoptysis, and dyspnea) and side-effects from chemo- and radiotherapy (e.g., hair loss, neuropathy, sore mouth and dysphagia). With the exception of 2 pain questions, which have dichotomous response categories (no or yes) and a free response if 'yes' is selected, all items on the QLQ-LC13 are scored on a 4-point Likert scale ranging from 1 (not at all) to (very much). The items have a 1-week recall period. All scale and item scores are linearly transformed to a 0 to 100 scale, with higher scores representing increasing symptom levels or impacts.
Change in Physical Functioning using EORTC QLQ-LC13 in the Overall Population | Up to 41 Months
  The EORTC QLQ-LC13 is the lung cancer specific module of the core EORTC QLQ-C30.2 The QLQ-LC13 includes 13 questions that include both multi-item and single-item scales of lung cancer-associated symptoms (e.g., pain, coughing, hemoptysis, and dyspnea) and side-effects from chemo- and radiotherapy (e.g., hair loss, neuropathy, sore mouth and dysphagia). With the exception of 2 pain questions, which have dichotomous response categories (no or yes) and a free response if 'yes' is selected, all items on the QLQ-LC13 are scored on a 4-point Likert scale ranging from 1 (not at all) to (very much). The items have a 1-week recall period. All scale and item scores are linearly transformed to a 0 to 100 scale, with higher scores representing increasing symptom levels or impacts.
Change in Physical Functioning as Measured by the Physical Functioning Domain of the EORTC QLQ-C30 in the Population of Participants with no CNS Metastases at Baseline | Up to 41 Months
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.
Change in Physical Functioning as Measured by the Physical Functioning Domain of the EORTC QLQ-C30 in the Overall Population | Up to 41 Months
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.
Change in Quality of Life as Measured by the Global Health Status/Quality of Life Domain of the EORTC QLQ-C30 in the Population of Participants with no CNS Metastases at Baseline | Up to 41 Months
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.
Change in Quality of Life as Measured by the Global Health Status/Quality of Life Domain of the EORTC QLQ-C30 in the Overall Population | Up to 41 Months
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.
Percentage of Participants With Adverse Events (AEs) | Up to 41 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-142